CLINICAL TRIAL: NCT07168148
Title: Steroid Treatment for Elimination of Rebound Obstruction From Intranasal Decongestants
Acronym: STEROID
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202501224
Record Dates: First submitted 2025-05-29; First posted 2025-09-11 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Nasal Obstruction; Chronic Rhinitis
Keywords: topical intranasal corticosteroid management; nasal airway evaluation; triamcinolone; oxymetazoline
MeSH Terms: conditions — Nasal Obstruction | interventions — Oxymetazoline; Triamcinolone

STUDY DESIGN:
Intervention Model Description: prospective virtually administered
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Titration (Experimental): Participants will begin the trial by providing their average daily usage of oxymetazoline.
  They will then be stratified according to this usage and placed into a titration schedule. After a week on a given titration level, they will be assessed for severity of nasal obstruction and, if controlled, they will progress to the next lower titration level.
  Participants with twice daily use, will then be placed in a titration schedule for oxymetazoline concentration which will stop when the oxymetazoline concentration is set to zero.
  Interventions: Drug: Oxymetazoline + Triamcinolone

INTERVENTIONS:
Drug: Oxymetazoline + Triamcinolone — Participants will be stratified according to this usage and placed into a titration schedule.
  * Titration 1: 0.05% 5x/day,
  * Titration 2: 0.05% 4x/day,
  * Titration 3: 0.05 3x/day,
  * Titration 4: 0.05% 2x/day.
  Participants with twice daily use, will then be placed in a titration schedule for oxymetazoline concentration which will stop when the oxymetazoline concentration is set to zero.
  * Titration 5: 0.0375% Afrin/Nasacort 2x/day,
  * Titration 6: 0.025% Afrin/Nasacort 2x/day,
  * Titration 7: 0.0125% Afrin/Nasacort 2x/day,
  * Titration 8: 0.0% Afrin/Nasacort 2x/day.
  Other Names: Afrin + Nasacort

SUMMARY:
This prospective, virtually administered trial conducted throughout the United States aims to evaluate a standardized protocol including the serial dilution of topical decongestants with concurrent topical steroids (triamcinolone), for elimination of dependence on topical decongestants.

DETAILED DESCRIPTION:
Participants will begin the trial by providing their average daily usage of oxymetazoline. They will then be stratified according to this usage and will be placed into a titration schedule. In the first week of the trial they will continue their usage of oxymetazoline plus twice daily triamcinolone intranasal spray. Continuing twice daily triamcinolone intranasal spray, the oxymetazoline dosage will be decreased each week until it matches the triamcinolone frequency. Each week following this point the subjects will continue with a mixture of different concentrations of oxymetazoline till complete elimination.

The maximum treatment time for participants who start the trial in the highest frequency oxymetazoline use group (greater than or equal to 5 times per day) would be 8 weeks.

After a week on a given titration level, they will be assessed for severity of nasal obstruction and, if controlled, they will progress to the next titration.

ELIGIBILITY:
Inclusion Criteria:

2) have a history of chronic nasal obstruction 3) at least daily topical decongestant usage for at least 3 months 4) ability to read, write, and understand English.

Exclusion Criteria:

1. Any history of sinonasal mass/tumor
2. Any history of nasal polyps
3. Septal perforation
4. A diagnosis of one of the following conditions:

   1. eosinophilic granulomatosis with polyangiitis
   2. granulomatosis with polyangiitis
5. Any current intranasal drug use such as cocaine.
6. If they are currently using or have used intranasal steroid medications (oral or nasal) besides oxymetazoline for the past month.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-11-10 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Responder rate | week 8
  The primary outcome measure will be the responder rate, defined as the percentage of participants who are able to discontinue decongestant use by the end of the study period and report that their symptoms are well-controlled, indicated by a score of 4 or less on the CGI-S.

SECONDARY OUTCOMES:
Responder rate among supratherapeutic users. | week 8
  Responder rate among supratherapeutic users, will be defined as percentage of participants who started the study using topical decongestants more than twice per day and who are able to discontinue decongestant use by the end of the study period and report that their symptoms are well-controlled, indicated by a score of 4 or less on the CGI-S.
The rate of partial responders among supratherapeutic users | week 8
  The rate of partial responders among supratherapeutic users will be defined as the percentage of supratherapeutic users who achieve a reduction in their usage of decongestants to twice daily by the end of the study.
Change in Nasal Obstruction Symptom Evaluation (NOSE) | through study completion, on average of 8 weeks
  NOSE is a disease-specific survey designed to measure nasal obstruction. It consists of 5 questions, each rated on a scale of 0 to 4, and the total score represents the sum of the raw scores multiplied by 5. A score of 30 is considered indicative of clinically significant NAO.
  Change in Nasal Obstruction Symptom Evaluation (NOSE) will be calculated as the difference in NOSE score at baseline minus NOSE score at the end of study participation.

CONTACTS AND LOCATIONS:
Overall Officials: Nyssa Farrell, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Settipane RA, Charnock DR. Epidemiology of rhinitis: allergic and nonallergic. Clin Allergy Immunol. 2007;19:23-34. PMID 17153005
- [Background] Mehuys E, Gevaert P, Brusselle G, Van Hees T, Adriaens E, Christiaens T, Van Bortel L, Van Tongelen I, Remon JP, Boussery K. Self-medication in persistent rhinitis: overuse of decongestants in half of the patients. J Allergy Clin Immunol Pract. 2014 May-Jun;2(3):313-9. doi: 10.1016/j.jaip.2014.01.009. Epub 2014 Mar 29. PMID 24811023
- [Background] LAKE CF. Rhinitis medicamentosa. Proc Staff Meet Mayo Clin. 1946 Sep 18;21(19):367-71. No abstract available. PMID 20274226
- [Background] Feinberg AR, Feinberg SM. The "nose drop nose" due to oxymetazoline (Afrin) and other topical vasoconstrictors. IMJ Ill Med J. 1971 Jul;140(1):50-2. No abstract available. PMID 4104967
- [Background] Hallen H, Enerdal J, Graf P. Fluticasone propionate nasal spray is more effective and has a faster onset of action than placebo in treatment of rhinitis medicamentosa. Clin Exp Allergy. 1997 May;27(5):552-8. PMID 9179430
- [Background] Ferguson BJ, Paramaesvaran S, Rubinstein E. A study of the effect of nasal steroid sprays in perennial allergic rhinitis patients with rhinitis medicamentosa. Otolaryngol Head Neck Surg. 2001 Sep;125(3):253-60. doi: 10.1067/mhn.2001.117717. PMID 11555762
- [Background] Scadding GK. Rhinitis medicamentosa. Clin Exp Allergy. 1995 May;25(5):391-4. doi: 10.1111/j.1365-2222.1995.tb01068.x. No abstract available. PMID 7553240
- [Background] Vaidyanathan S, Williamson P, Clearie K, Khan F, Lipworth B. Fluticasone reverses oxymetazoline-induced tachyphylaxis of response and rebound congestion. Am J Respir Crit Care Med. 2010 Jul 1;182(1):19-24. doi: 10.1164/rccm.200911-1701OC. Epub 2010 Mar 4. PMID 20203244
- [Background] Graedon, Terry. "How to Beat Nose Spray Dependence One Nostril at a Time." Https://Www.Peoplespharmacy.Com/, The People's Pharmacy, 27 Mar. 2023, www.peoplespharmacy.com/articles/how-to-beat-nose-spray-dependence-one- nostril-at-a-time.
- [Background] Afrin Addicts. [ca. 2024]. In Facebook [Group page]. Retrieved September 4, 2024, from https://www.facebook.com/groups/1551311815137595
- [Background] Park SSE, Barmettler A. Vision Loss Secondary to Facial and Periorbital Steroid Injection: A Systematic Review. Ophthalmic Plast Reconstr Surg. 2021 Nov-Dec 01;37(6):511-521. doi: 10.1097/IOP.0000000000001910. PMID 33481540
- [Background] Elwany SS, Stephanos WM. Rhinitis medicamentosa. An experimental histopathological and histochemical study. ORL J Otorhinolaryngol Relat Spec. 1983;45(4):187-94. doi: 10.1159/000275642. PMID 6192384
- [Background] Elwany S, Abdel-Salaam S. Treatment of rhinitis medicamentosa with fluticasone propionate--an experimental study. Eur Arch Otorhinolaryngol. 2001 Mar;258(3):116-9. doi: 10.1007/s004050000309. PMID 11374251
- [Background] Knipping S, Holzhausen HJ, Goetze G, Riederer A, Bloching MB. Rhinitis medicamentosa: electron microscopic changes of human nasal mucosa. Otolaryngol Head Neck Surg. 2007 Jan;136(1):57-61. doi: 10.1016/j.otohns.2006.08.025. PMID 17210334
- [Background] Lin CY, Cheng PH, Fang SY. Mucosal changes in rhinitis medicamentosa. Ann Otol Rhinol Laryngol. 2004 Feb;113(2):147-51. doi: 10.1177/000348940411300213. PMID 14994772
- [Background] Cam B, Sari M, Midi A, Gergin O. Xylitol treats nasal mucosa in rhinitis medicamentosa: an experimental rat model study. Eur Arch Otorhinolaryngol. 2019 Nov;276(11):3123-3130. doi: 10.1007/s00405-019-05605-3. Epub 2019 Aug 29. PMID 31468129
- [Background] Suh SH, Chon KM, Min YG, Jeong CH, Hong SH. Effects of topical nasal decongestants on histology of nasal respiratory mucosa in rabbits. Acta Otolaryngol. 1995 Sep;115(5):664-71. doi: 10.3109/00016489509139384. PMID 8928640
- [Background] Tas A, Yagiz R, Yalcin O, Uzun C, Huseyinova G, Adali MK, Karasalihoglu AR. Use of mometasone furoate aqueous nasal spray in the treatment of rhinitis medicamentosa: an experimental study. Otolaryngol Head Neck Surg. 2005 Apr;132(4):608-12. doi: 10.1016/j.otohns.2005.01.010. PMID 15806055
- [Background] Busner J, Targum SD. The clinical global impressions scale: applying a research tool in clinical practice. Psychiatry (Edgmont). 2007 Jul;4(7):28-37. PMID 20526405
- [Background] Lipan MJ, Most SP. Development of a severity classification system for subjective nasal obstruction. JAMA Facial Plast Surg. 2013 Sep-Oct;15(5):358-61. doi: 10.1001/jamafacial.2013.344. PMID 23846399
- [Result] Graf P. Rhinitis medicamentosa: a review of causes and treatment. Treat Respir Med. 2005;4(1):21-9. doi: 10.2165/00151829-200504010-00003. PMID 15725047